CLINICAL TRIAL: NCT00853346
Title: Psychosocial Treatment of Depression in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Amy Farabaugh, PhD (Other)
Collaborators: Brigham and Women's Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Sponsor-Investigator, Amy Farabaugh, PhD, Director, Psychotherapy Research, Depression Clinical & Research Program, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MH076037-01
Record Dates: First submitted 2009-02-27; First posted 2009-03-02 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-11

CONDITIONS: Major Depressive Disorder; Parkinson's Disease
Keywords: Depression; Parkinson's Disease; Major Depression; Cognitive Behavioral Therapy
MeSH Terms: conditions — Depressive Disorder, Major; Parkinson Disease; Depression | interventions — Cognitive Behavioral Therapy; Therapeutics; Psychosocial Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients randomized to the immediate arm will be given 12 weeks of CBT starting one week after randomization
  Interventions: Behavioral: Cognitive Behavioral Therapy
- 2 (Active Comparator): Patients in the delayed arm will receive 12 weeks of CBT, starting 12 weeks after randomization.
  Interventions: Behavioral: Cognitive Behavioral Therapy

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy — 12 weeks of Cognitive Behavioral Therapy designed for adults with Parkinson's Disease and comorbid Depression
  Other Names: CBT; Cognitive Therapy; Therapy; Psychosocial Intervention
  Arms: 1
Behavioral: Cognitive Behavioral Therapy — 12 weeks of Cognitive Behavioral Therapy designed for adults with Parkinson's Disease and comorbid Depression
  Other Names: CBT; Cognitive Therapy; Therapy; Psychosocial Intervention
  Arms: 2

SUMMARY:
The purpose of the study is to examine the effects of a form of talk therapy called cognitive behavior therapy (CBT) in the treatment of major depression in individuals with Parkinson's disease (PD).

DETAILED DESCRIPTION:
CBT is a specific type of treatment that has been shown to be as helpful in treating depression as medications for depression. CBT focuses on thoughts, feelings, and behaviors. It focuses on the here and now, rather than the past. CBT offers concrete strategies and skills for coping with depression, PD, and other life problems. Previous research leads us to believe that this type of therapy may help people with PD cope with their depression.

ELIGIBILITY:
Inclusion Criteria:

In addition to the DSM-IV diagnostic criteria for major depressive disorder, the following conditions must be met for patient eligibility:

* Written informed consent.
* Subjects with a primary diagnosis of PD who also currently meet DSM-IV criteria for MDD
* Subjects must be stable on their anti-Parkinson treatment, as defined by no medication changes over the past 6 weeks
* Subjects may be taking an antidepressant as long as they have had a stable dose for up to 6 weeks and do not alter the dosage during the course of the study
* Men or women 40-80 years of age
* HAMD-17 scores > 14 at screen visit
* Score of 25 or greater on the Mini-Mental Status Examination
* Willing to come to MGH for screening and study participation

Exclusion Criteria:

Patients meeting any of the following criteria are to be excluded from the study:

* Subjects who, in the investigator's judgment, pose a current, serious suicidal or homicidal risk
* Patients who would not be appropriate for a delayed CBT control due to the severity of their depression based on clinical judgment as well as HAMD-17 scores > 28
* The following DSM-IV diagnoses: 1) substance use disorders, including alcohol dependence, active within the last 3 months; 2) schizophrenia; 3) delusional disorder; 4) psychotic disorders not elsewhere classified; 5) bipolar disorder; 6) MDD with psychotic features
* Subjects who meet DSM-IV criteria for dementia
* Severe, unstable concurrent medical conditions (determined by his/her physician) that are likely to require hospitalization within six months from study entry (e.g., a patient with severe congestive heart failure who has a history of recent hospital admissions)
* Subjects may not be receiving a psychosocial intervention that is specific for depression; psychosocial interventions not specific for depression (e.g., couples counseling) and established for three or more months before screen visit are allowed

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2007-04; Primary Completion 2013-04 (Estimated); Study Completion 2013-04 (Estimated)

PRIMARY OUTCOMES:
Response according to the Hamilton Rating Scale for Depression, 17 items (HAM-D 17). | screen, week 4, week 8, week 12; if applicable, week 16, week 20, week 24

CONTACTS AND LOCATIONS:
Overall Officials: Amy Farabaugh, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States